CLINICAL TRIAL: NCT05854472
Title: The Effect of a Smartphone Application Developed for Patients With Liver Transplantation on Adherence to Immunosuppressive Drug Use, Anxiety and Quality of Life: Randomized Controlled Trial
Brief Title: Using Smartphone Application After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sbu-asavsar-hayhan-001
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2023-02

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; drug adherence; quality of life; anxiety; smartphone application
MeSH Terms: conditions — Medication Adherence; Anxiety Disorders

STUDY DESIGN:
Masking Description: there is no masking in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of smartphone application (Experimental): A smartphone application content will be developed to facilitate the use of immunosuppressive drugs by individuals with liver transplantation and to provide guidance to patients. The effect of smartphone application usage on immunosuppressive drug compliance, anxiety and quality of life in liver transplant patients will be evaluated.
  Interventions: Other: smartphone based application use
- not use a smart phone application (No Intervention): In this group, patients who have liver transplantation and do not use a smart phone application for liver transplantation patients after discharge will be included.

INTERVENTIONS:
Other: smartphone based application use — A smartphone application content will be developed to facilitate the use of immunosuppressive drugs by individuals with liver transplantation and to provide guidance to patients. The effect of smartphone application usage on immunosuppressive drug compliance, anxiety and quality of life in liver transplant patients will be evaluated.
  Arms: Use of smartphone application

SUMMARY:
The aim of this randomized controlled clinical study was a study that could facilitate the management of immunosuppressive therapy, including information specific to liver transplant patients, to increase immunosuppressive medication adherence and quality of life, and reduce anxiety in the early period in patients who have to use lifelong immunosuppressive medication to prevent organ rejection after liver transplantation. The aim of this study is to develop a smartphone application and evaluate the effectiveness of the application.

Research Question: What is the effect of smartphone application use on immunosuppressive medication adherence, anxiety and quality of life in patients undergoing liver transplant?

Research Hypotheses

H11: There is a difference between medication adherence in patients who use and do not use smartphone applications after liver transplantation at the 3rd month after discharge.

H21: There is a difference between the anxiety levels of the patients who used and did not use smart phone applications after liver transplantation in the first month after discharge.

H31: There is a difference between the anxiety levels of the patients using and not using smart phone applications after liver transplantation at the 3rd month after discharge.

H41: There is a difference between the quality of life of patients using and not using a smart phone application after liver transplantation, at the first month after discharge.

H51: There is a difference between the quality of life of patients who use and do not use smart phone applications after liver transplantation at the 3rd month after discharge.

H61: There is a difference between immunosuppressive blood drug levels in the 1st month after discharge in patients who use and do not use smart phone applications after liver transplantation.

H71: There is a difference between the immunosuppressive blood drug levels in the 3rd month after the discharge of the patients who used and did not use the smart phone application after liver transplantation.

H81: There is a difference between the rejection rates of patients who use and do not use smartphone applications after liver transplantation, within the 3 months after hospital discharge.

H91: There is a difference between the rates of readmission within the 3 months after hospital discharge in patients who use and do not use smart phone applications after liver transplantation.

Researchers will compare the experimental and control groups to see if there is a difference between patients' adherence to medication, quality of life, and anxiety levels. The experimental group is going to use the smartphone application developed specifically for patients with liver transplantation for 3 months.

DETAILED DESCRIPTION:
During the lifelong immunosuppressive treatment after liver transplantation and in the process of adapting to this treatment, patients may experience difficulties in compliance with drug use. For this reason, the quality of life of patients is affected and psychiatric problems may occur. When studies on improving adherence to immunosuppressive therapy and improving quality of life after solid organ transplantation were examined, it was observed that interventional studies in the liver population were insufficient. The aim of this project, which is planned in this direction, is a smart phone application that contains information specific to liver transplantation patients in order to increase medication adherence and quality of life and reduce anxiety in the early period in patients who have to use lifelong immunosuppressive drugs to prevent organ rejection after liver transplantation. The aim of this study is to develop a smartphone application and evaluate the effectiveness of the application.

In the content of the smartphone application;

* Time of drug use, reminder of the dose to be taken, drug information, drug-drug interactions and drug-food interactions information,
* Patients' blood pressure, blood glucose values, immunosuppressive blood level
* Patients can record and/or review the side effects, and take their own notes on the application, such as the subjects they want to convey to their doctor when they go to follow-up and controls,
* Information about liver transplantation and life after it,
* Reminding the appointment time,
* Individual counseling (Patients leave questions to the researcher via the application on the subjects they need),
* The interaction of the drugs used with the environmental factor (the effect of the air temperature in the city on the patient),
* Notices encouraging a healthy lifestyle (drinking water, walking, exercising, not smoking, not drinking alcohol, etc.),

This study was planned as a single-center, randomized controlled clinical trial. Study sample; by taking 5% margin of error (α = 0.05) and 80% power (1-β = 0.80), the number of samples for each group was calculated as 23, a total of 46. Due to possible data loss, it is aimed to reach 60 patients, 30 in each group. In this project, a practical smartphone application will be developed that will meet the needs of patients undergoing liver transplantation and that they can easily carry with them.

In data collection, "Patient Description and Clinical Characteristics Form", "Immunosuppressive Treatment Adherence Scale", "Immunosuppressive Drug Adherence Scale", "Hospital Anxiety and Depression Scale", "SF-36 Quality of Life Scale", "Turkish-Computer System Usability Questionnaire Short Version Scale" and patients' immunosuppressive blood drug levels from hospital records will be used. Data were collected before patients were discharged, at 1 month postoperatively, and at 3 months postoperatively.

When parametric test prerequisites are met in the analysis of the data; It is envisaged to use Chi-Square Test, Mc Neamer test, Independent Sample T Test, Pearson Correlation Analysis, Analysis of Variance in Repeated Measurements, Bonferroni test as multiple comparison method. If the parametric test prerequisites are not met, it is predicted that Mann Whitney U test, Wilcoxon Test, Friedman Test and Spearman Correlation Analysis will be used.

The results of this study show that a new practical application, in which patients can follow the importance, effect, side effects and dose and hours of immunosuppressive drugs, in the difficult process that needs to be struggled with compliance with immunosuppressive drug hours after liver transplantation, fear of organ rejection and immunosuppressive treatment side effects, will help to improve drug compliance. It is predicted that it will reduce anxiety about drug treatment in the early period and increase the quality of life of the patient by increasing the patient's quality of life. In addition, it is thought that increasing drug compliance will reduce re-hospitalizations and organ rejection.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* First time liver transplant and planning of discharge
* Using at least one immunosuppressive drug
* Ability to use immunosuppressive drugs independently
* Absence of mental and auditory disabilities
* Absence of a psychiatric disorder and not using drugs
* No problem in speaking and understanding Turkish
* Using a smartphone for at least 6 months
* Being an Android smartphone user
* Having an internet connection
* Agreeing to participate in the research voluntarily

Exclusion Criteria:

* Failure to communicate with the patient before the data collection phases are over.
* Leaving work voluntarily
* Development of organ rejection during the data collection phase
* The patient's death during the data collection phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 3 months
  Two different scales called Immunosuppressive Treatment Adherence Scale (4 items) and Immunosuppressive Medication Adherence Scale (11 items) will be used to determine the medication adherence reported by the patients after 3 months of discharge. As a result of the Immunosuppressive Treatment Adherence Scale, the lowest 0 and the highest 12 points are obtained. 0 indicates very poor compliance and 12 indicates excellent compliance. On the Scale of Adherence to Drug Use, the lowest score is 11 and the highest score is 55. The increase in the score obtained from the scale indicates that the individual's compliance with the use of immunosuppressive drugs increases.
the blood level of the immunosuppressive drug | 1month
  In order to determine the drug compliance of the patients, the blood level of the immunosuppressive drug will be checked in 1 month after discharge. Tacrolimus normal level will be evaluated according to the reference range of 5-15 mg/dl in the hospital protocol where the study will be conducted. The fact that the blood drug level is outside the reference range will be considered as an indicator of the patient's low compliance with the use of immunosuppressive drugs.
the blood level of the immunosuppressive drug | 3 months
  In order to determine the drug compliance of the patients, the blood level of the immunosuppressive drug will be checked in 3 months after discharge. Tacrolimus normal level will be evaluated according to the reference range of 5-15 mg/dl in the hospital protocol where the study will be conducted. The fact that the blood drug level is outside the reference range will be considered as an indicator of the patient's low compliance with the use of immunosuppressive drugs.

SECONDARY OUTCOMES:
Anxiety Levels | 1 month
  After 1 month after discharge, patients will complete the 14-item Hospital Anxiety and Depression Scale to determine the patients' anxiety status. The cut-off points for the Hospital Anxiety and Depression Scale are 10 for the anxiety subscale and 7 for the depression subscale. Patients with scores above these scores can be considered as a risk group.
Anxiety Levels | 3 months
  After 3 months after discharge, patients will complete the 14-item Hospital Anxiety and Depression Scale to determine the patients' anxiety status. The cut-off points for the Hospital Anxiety and Depression Scale are 10 for the anxiety subscale and 7 for the depression subscale. Patients with scores above these scores can be considered as a risk group.Odd-numbered items in the scale are anxiety, and even-numbered items are depression.In this study, the anxiety subscale of the scale will be used.
Life Quality | 1 month
  After spending 1 month after discharge, patients will complete the SF-36 Quality of Life Scale, which consists of 36 items, to evaluate the patients' quality of life levels. The scale with a positive score was scored so that the higher the score of each health area, the higher the health-related quality of life.
Life Quality | 3 months
  After spending 3 months after discharge, patients will complete the SF-36 Quality of Life Scale, which consists of 36 items, to evaluate the patients' quality of life levels. The scale with a positive score was scored so that the higher the score of each health area, the higher the health-related quality of life.
Rejection rates | 3 months
  Rejection rates are going to be collected from hospital records by the researchers. The high rates will be associated with the non-compliance of the patients to their drug use.
Readmission Rates | 3 months
  Readmission rates are going to be collected from hospital records by the researchers. The high rates will be associated with the non-compliance of the patients to their drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faust A, Stine JG. Leveraging the Coronavirus Disease 2019 Pandemic: Is It Time to Consider Incorporating Mobile Applications Into Standard Clinical Management of the Liver Transplantation Patient? Liver Transpl. 2021 Apr;27(4):479-481. doi: 10.1002/lt.25991. Epub 2021 Mar 5. No abstract available. PMID 33484229
- [Background] Dobbels F, De Bleser L, Berben L, Kristanto P, Dupont L, Nevens F, Vanhaecke J, Verleden G, De Geest S. Efficacy of a medication adherence enhancing intervention in transplantation: The MAESTRO-Tx trial. J Heart Lung Transplant. 2017 May;36(5):499-508. doi: 10.1016/j.healun.2017.01.007. Epub 2017 Jan 6. PMID 28162931
- [Background] Harrison JJ, Badr S, Hamandi B, Kim SJ. Randomized Controlled Trial of a Computer-Based Education Program in the Home for Solid Organ Transplant Recipients: Impact on Medication Knowledge, Satisfaction, and Adherence. Transplantation. 2017 Jun;101(6):1336-1343. doi: 10.1097/TP.0000000000001279. PMID 27367473